CLINICAL TRIAL: NCT05296356
Title: OSU6162 in Bipolar Depression: An Open-label, Flexible Dose Study (OBID)
Brief Title: OSU6162 in Bipolar Depression (OBID)
Acronym: OBID
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Arvid Carlsson Research AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT number: 2020-001980-95; 2024-517560-30-00 (EU CTIS Number); 2020-001980-95 (EudraCT Number)
Record Dates: First submitted 2021-11-08; First posted 2022-03-25 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Bipolar Depression
MeSH Terms: conditions — Bipolar Disorder | interventions — OSU 6162

STUDY DESIGN:
Intervention Model Description: Open study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OSU6162 (Experimental): Coated tablet, flexible dosing
  Interventions: Drug: OSU6162

INTERVENTIONS:
Drug: OSU6162 — OSU6162

SUMMARY:
An explorative, open label, single armed, flexible dose, single center, phase IIa study of 8 weeks, initiated in subjects with bipolar depression. The study will consist of 9 visits and 1 safety visit.

Subjects with a primary diagnosis of bipolar disorder (type 1 or 2) currently in an acute depressive phase (i.e. bipolar depression) and being on stable medication with at least one mood stabilizer.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Voluntary admission to the psychiatric ward prior or directly after the screening point
3. Age: 18-65 on the day of screening
4. Meeting DSM-5 criteria for a depressive episode in Bipolar Disorder type I or type II, as confirmed by the Mini International Neuropsychiatric Interview (MINI)
5. Displaying a sum score of ≥10 on the Bech 6-item subscale of the Hamilton Depression rating Scale.
6. Treatment with a stable dose of a mood stabilizer since at least 4 weeks before screening: lithium s-conc> 0,45 mmol/L; >lamotrigine dose 100 mg/d; >valproate dose > 900 mg/d, >carbamazepine concentration >20 mmol/L
7. In female patients of childbearing potential: negative result of a pregnancy test and a method of contraception with a failure rate of less than 1 %. Women of childbearing potential must, for inclusion, use a highly efficient method of contraception, i.e. a method with a failure rate of less than 1% (e.g. sterilization, hormone implants, hormone injections, some intrauterine devices, or vasectomy in partner).
8. Male patients must agree to use condoms during the study and for 2 weeks after the end of the study/last dose of IMP, unless their partner is using a highly efficient method of contraception, as described above.

Exclusion Criteria:

1. Ongoing compulsory care.
2. Subject is considered by the investigator to be at imminent risk of suicide or injury to self, others, or property.
3. Previously diagnosed or meeting MINI criteria at interview for obsessive-compulsive disorder or post-traumatic stress disorder.
4. A previous diagnosis of a personality disorder, autism, ADHD, or intellectual disability.
5. A history of substance/alcohol abuse within 2 years prior to screening.
6. Any other previously diagnosed or suspected CNS disorder that according to the investigator renders the patient unsuitable for participation in the trial (such as dementia, brain injury, and epilepsy).
7. Young Mania Rating Scale (YMRS) total score of >12 at screening or at any time during the trial.
8. Any somatic illness that according to the investigator renders the patient unsuitable for participation in the trial.
9. Any signs or symptoms of somatic illness resulting from assessment of vital signs, physical examination, clinical laboratory tests or 12- lead ECG that according to the investigator renders the patient unsuitable for participation for safety reasons, including a QTc-time on ECG exceeding 450 ms in men and 460 ms in women.
10. Any factor that according to the investigator renders it unlikely that the patient will comply with the instructions regarding treatment, visits etc.
11. Any change in medication (including dosage) of an antidepressant drug or a mood stabiliser within 4 weeks prior to screening or at any time during the trial.
12. Ongoing treatment with potent cytochrome P450 enzyme inhibitors (e.g., bupropion, fluvoxamin, ketoconazol, itraconazole, telitromycin, clarithromycin, protease inhibitors, quinidine, and terbinafine).
13. Ongoing treatment with drugs displaying a narrow therapeutic window - with the exception of lithium - where either reduced or increased serum levels are potentially harmful (including but not limited to warfarin, other anticoagulants, digoxin. other antiarrythmics, anticonvulsants when prescribed for treatment of epilepsy but not when prescribed for bipolar disorder, cyclosporine, and immunosuppressants).
14. Ongoing treatment with drugs with dopaminergic synapses as primary site of action (e.g., antipsychotics, bupropion, central stimulants, and drugs for Parkinson's disease).
15. No observed beneficial effect of treatment and a symptom severity that by the investigator's assessment would render continued participation unethical.
16. Previous intake of OSU6162.
17. Current participation in another clinical trial.
18. Nursing women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2021-10-25 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the Montgomery-Åsberg Depression Rating Scale (MADRS) at endpoint [Day 60]. | Endpoint at 60 days treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Sahlgrenska university hospital/Östra, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No